CLINICAL TRIAL: NCT04863014
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Evinacumab in Patients With Severe Hypertriglyceridemia for the Prevention of Recurrent Acute Pancreatitis
Brief Title: Efficacy and Safety of Evinacumab in Adult Patients With Severe Hypertriglyceridemia for the Prevention of Recurrent Acute Pancreatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1500-HTG-20118; 2021-000437-13 (EudraCT Number)
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hypertriglyceridemia
Keywords: Severe Hypertriglyceridemia (HTG); Recurrent Acute Pancreatitis
MeSH Terms: conditions — Hypertriglyceridemia; Pancreatitis | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- evinacumab (Experimental): Randomized 1:1
  Interventions: Drug: evinacumab
- Placebo (Placebo Comparator): Randomized 1:1
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: evinacumab — Intravenous infusion every 4 weeks (Q4W)
  Other Names: REGN1500; Evkeeza™
  Arms: evinacumab
Other: Placebo — Intravenous infusion Q4W
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the proportion of patients with elevated triglycerides (TG), without familial chylomicronemia syndrome (FCS) due to loss of function (LoF) mutations in lipoprotein lipase (LPL), and a history of hypertriglyceridemia (HTG)-associated acute pancreatitis (AP) who experience a recurrent episode of AP after treatment with evinacumab versus placebo.

The secondary objectives of the study are:

* To determine the change in the standard lipid profile after therapy with evinacumab versus placebo
* To determine the changes in specialty lipoprotein parameters (ApoC3, ApoB48, ApoB100, and nuclear magnetic resonance [NMR] lipid profile) after therapy with evinacumab versus placebo
* To measure the number of AP episodes per patient
* To assess the safety and tolerability of evinacumab
* To assess the potential immunogenicity of evinacumab
* To assess the concentrations of total evinacumab and total angiopoietin-like 3 (ANGPTL3)

ELIGIBILITY:
Key Inclusion Criteria:

1. Adults without FCS due to LPL loss of function mutations
2. Documented history of 1 HTG-associated AP episode within 24 months of screening
3. Fasting serum TG value >880 mg/dL (10 mmol/L) or >500 mg/dL (5.6mmol/L) determined during the screening period as described in the protocol
4. Stable dose of lipid-lowering therapy (≥8 weeks) and willingness to maintain a stable regimen throughout the study
5. Body mass index ≥18.0 and ≤45.0 kg/m2
6. Compliance with a stable diet and exercise regimen at screening and willingness to continue the diet through the end of the study

Key Exclusion Criteria:

1. Hospitalization for AP within 4 weeks of screening
2. Known genetic FCS defined as homozygous or compound heterozygous LoF mutations in LPL as defined in the protocol
3. Symptomatic gallstone disease within 6 months prior to screening as defined in the protocol
4. Use of any medication or nutraceutical known to alter serum lipids which has not been part of a stable therapeutic regimen for at least 8 weeks, and there are no plans to change the regimen during the study
5. Presence of any clinically significant, uncontrolled endocrine disease known to influence serum lipids as defined in the protocol
6. Has received a COVID-19 vaccination within 1-week of planned start medication or for which the planned COVID-19 vaccination would not be completed 1-week prior to start of the study

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (39):
- United States (32):
  - Radin Cardivascular Medical Group, Inc, Newport Beach, California
  - Yale Cancer Center - Yale University, New Haven, Connecticut
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Harmony Medical Research Institute, Inc., Hialeah, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - NorthShore Medical Group, Evanston, Illinois
  - Advocate Medical Group Midwest Heart Specialists, Park Ridge, Illinois
  - Methodist Medical Center of Illiniois - UnityPoint Clinic, Peoria, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - St. Vincent Medical Group, Inc., Carmel, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health, Manhasset, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Weill Cornell Medical College, New York, New York
  - Mt Sinai - Ichan Medical Institute, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Methodist Dallas Medical Center, Dallas, Texas
  - Sante Clinical Research, Kerrville, Texas
  - University of Washington, Seattle, Washington
  - MultiCare Institute for Research, Spokane, Washington
  - West Virginia University Heart & Vascular Institute, Morgantown, West Virginia
  - Wisconsin Center for Advanced Research - a division of GI Associates, LLC, Milwaukee, Wisconsin
- Canada (3):
  - Robarts Research Institute, London, Ontario
  - Centre Etudes Cliniques Ecogene-21, Chicoutimi, Quebec
  - Clinique des maladies lipidiques de Quebec, Québec
- Germany (2):
  - University Hospital Carl Gustav Carus, Dresden
  - University Hospital of Leipzig, Leipzig
- Netherlands (2):
  - Amsterdam University Medical Center (Amsterdam UMC), Academic Medical Center (AMC), Amsterdam
  - Ziekenhuis Rijnstate, Arnhem

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 40 participants were screened, of which 21 participants met the eligibility criteria and were randomized in 1:1 to receive either evinacumab or matched placebo. The sponsor terminated the study early due to enrollment issues.
Groups:
- Evinacumab: Participants received evinacumab 20 milligrams per kilogram (mg/kg) IV infusion Q4W starting from Day 1 up to 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Evinacumab
Started | 10 | 11
Completed | 7 | 5
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Subject Decision | 0 | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) included all participants who received at least 1 dose or part of a dose of double-blind study drug.
Groups:
- Evinacumab: Participants received evinacumab 20 mg/kg IV infusion Q4W starting from Day 1 up to 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Evinacumab | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.0 (15.22) | 45.3 (9.46) | 45.6 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change in Apolipoprotein C3 (ApoC3) From Baseline to Week 52
Description: Apolipoproteins transport lipids through the body by binding with fat and cholesterol to form lipoproteins. ApoC3 was a component of very-low-density lipoproteins (VLDL), high-density lipoprotein (HDL), and triglyceride-rich chylomicrons and regulates lipid metabolism. Percent change in ApoC3 from Baseline to Week 52 was reported.
Time Frame: Baseline to week 52
Population: ITT population was defined as all randomized participants who received 1 dose or part of a dose of study drug. Here, "Overall number of participants analyzed" refers to participants who were evaluable for this outcome measure and "0" in the overall analyzed field signifies that none of the participants were available for the assessment at the specified timepoint for placebo arm.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Placebo: Randomized 1:1 Participants received matched-placebo IV infusion Q4W starting from Day 1 up to 52 weeks.
- Evinacumab: Randomized 1:1 Participants received evinacumab 20 mg/kg IV infusion Q4W starting from Day 1 up to 52 weeks.
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | -73.78

2. Secondary Outcome: Percent Change in Fasting Triglycerides (TGs) - (From Baseline to Week 52)
Time Frame: Baseline to week 52
Population: The ITT population is defined as all randomized participants who received 1 dose or part of a dose of study drug. Participants in the ITT population will be analyzed according to the treatment group allocated by randomization. Participants who were evaluable for this outcome measure and "0" in the overall analyzed field signifies that none of the participants were available for the assessment at the specified timepoint for placebo arm.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Evinacumab: Randomized 1:1 Randomized 1:1 Participants received evinacumab 20 mg/kg IV infusion Q4W starting from Day 1 up to 52 weeks.
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | -92.88

3. Secondary Outcome: Percent Change in Total Cholesterol (TC) - (Baseline to Week 52)
Time Frame: Baseline to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | -57.62

4. Secondary Outcome: Percent Change in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) - (From Baseline to Week 52)
Time Frame: Baseline to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | -60.12

5. Secondary Outcome: Percent Change in Apolipoprotein B48 (ApoB48) From Baseline to Week 52
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | -92.09

6. Secondary Outcome: Percent Change in Apolipoprotein B100 (ApoB100) Levels From Baseline to Week 52
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | 225.14

7. Secondary Outcome: Percent Change in Nuclear Magnetic Resonance (NMR)-Determined Particle Size and Number From Baseline to Week 52
Time Frame: Baseline to week 52
Population: Data was not collected and analyzed for this outcome measure as the sponsor terminated the study early due to enrollment issues.
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Independently Adjudicated Positive Episodes of Acute Pancreatitis (AP) Per Participant
Time Frame: Up to 52 weeks
Population: The ITT population is defined as all randomized participants who received 1 dose or part of a dose of study drug. Participants in the ITT population will be analyzed according to the treatment group allocated by randomization
Measure: Mean (Standard Deviation); unit: Number of Episodes
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 10 | 11
Number of Episodes | 0.1 (0.32) | 0.4 (0.67)

9. Primary Outcome: Percentage of Participants With at Least One Positively Adjudicated Acute Pancreatitis (AP) Episode
Description: All AP (Acute Pancreatitis) episodes occurred post-study drug treatment.
Time Frame: Baseline to 52 weeks
Population: The Intent-to-treat Analysis Set (ITT) population was defined as all randomized participants who received 1 dose or part of a dose of study drug.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: Participants received matched-placebo IV infusion Q4W starting from Day 1 up to 52 weeks.
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 10 | 11
Percentage of Participants | 10.0 | 27.3

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Time Frame: From start of study drug administration up to off drug follow-up (up to Week 72)
Population: The SAF included all participants who received at least 1 dose or part of a dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 10 | 11
Participants
  Participants with TEAEs | 10 | 7
  Participants with Serious TEAEs | 4 | 5

11. Secondary Outcome: Number of Participants With TEAEs Based on Severity
Description: AE was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. TEAEs are defined as AEs that developed or worsened during the treatment period. Severity of TEAEs was graded according to the following scale: Mild: Does not interfere in a significant manner with the participants normal functioning level, Moderate: Produces some impairment of functioning but is not hazardous to health and Severe: Produces significant impairment of functioning or incapacitation and is a definite hazard to the participants health.
Time Frame: From start of study drug administration up to off drug follow-up (up to Week 72)
Population: The SAF included all participants who received at least 1 dose or part of a dose of double-blind study drug. Here, "Overall number of participants analyzed" refers to participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 10 | 11
Participants
  Participants with Mild TEAEs | 3 | 3
  Participants with Moderate TEAEs | 3 | 1
  Participants with Severe TEAEs | 4 | 3

12. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Clinical laboratory parameters included biochemistry, hematology and urinalysis. The number of participants with clinically significant changes from baseline in laboratory parameters were reported. Clinical significance was determined by the investigator.
Time Frame: From start of study drug administration up to off drug follow-up (up to Week 72)
Population: The SAF included all participants who received at least 1 dose or part of a dose of double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Positive Treatment-emergent Anti-Drug Antibodies (ADA)
Description: Treatment-Emergent ADA was defined as any positive post baseline assay response when baseline results were negative or missing. Treatment-Emergent ADA responses were further classified as: Persistent (a positive result in the ADA assay detected in at least 2 consecutive post baseline samples separated by at least a 16-week post baseline period [based on] nominal sampling time], with no ADA-negative results in-between, regardless of any missing samples); Indeterminate (a positive result in the ADA assay at the last collection time point only, regardless of any missing samples); Transient (not persistent/indeterminate, regardless of any missing samples). Number of participants with positive treatment-emergent ADA response during Week 52 were reported.
Time Frame: Baseline to Week 52
Population: The ADA analysis set included all treated participants who received any amount of study drug (active or placebo) and had at least one non-missing ADA result following the first dose of the study drug or placebo. Here, "Overall number of participants analyzed" refers to participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 8 | 7
Participants
  Participants with Treatment-Emergent Response: Persistent | 0 | 0
  Participants with Treatment-Emergent Response: Transient | 0 | 0
  Participants with Treatment-Emergent Response: Indeterminate | 1 | 0

14. Secondary Outcome: Number of Participants With Positive Neutralizing Antibodies (NAb)
Description: NAb positive was defined as presence of at least one positive nAb sample.
Time Frame: Baseline to Week 52
Population: as for outcome 7
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percent Change in Fasting High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 52
Description: Percent Change in fasting HDL-C from Baseline to Week 52 was reported.
Time Frame: Baseline to Week 52
Population: The SAF included all participants who received at least 1 dose or part of a dose of double-blind study drug. Here, "Overall number of participants analyzed" refers to participants who were evaluable for this outcome measure and "0" in the overall analyzed field signifies that none of the participants were available for the assessment at the specified timepoint for placebo arm.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent change |  | 52.94

16. Secondary Outcome: Percent Change in Fasting Low Density Lipoprotein (LDL-C) From Baseline to Week 52
Description: LDL-C levels were determined in beta-quantification with ultracentrifugation method. Percent change in fasting LDL-C from Baseline to Week 52 was reported.
Time Frame: Baseline to Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 0 | 1
Percent Change |  | 695.00

17. Secondary Outcome: Concentration of Total Evinacumab in Serum
Description: Concentration of total evinacumab in serum by time at Pre-dose and End of Infusion were analyzed and reported.
Time Frame: Pre-dose and End of Infusion (EOI) at Weeks 0, 4, 8, 12, 16, 20, 24, 32, 36, 40, 44, and 48; Pre-dose at Weeks 28 and 52
Population: The PK analysis set included all randomized participants who received any study drug and for each participant who has at least 1 non-missing post-baseline measurement of evinacumab concentration. Here, "number analyzed" signifies to participants evaluable for this outcome at given timepoints. Data was planned to be reported only for evinacumab arm.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Evinacumab
Number analyzed (Participants) | 10
milligrams per liter (mg/L)
  Week 0: Pre-dose | 1.39 (4.40)
  Week 0: EOI (End of Infusion) | 573 (95.7)
  Week 4: Pre-dose: number analyzed (Participants) | 8
  Week 4: Pre-dose | 97.6 (37.4)
  Week 4: EOI (End of Infusion): number analyzed (Participants) | 8
  Week 4: EOI (End of Infusion) | 638 (286)
  Week 8: Pre-dose: number analyzed (Participants) | 8
  Week 8: Pre-dose | 133 (88.6)
  Week 8: EOI (End of Infusion): number analyzed (Participants) | 6
  Week 8: EOI (End of Infusion) | 724 (123)
  Week 12: Pre-dose: number analyzed (Participants) | 5
  Week 12: Pre-dose | 158 (81.1)
  Week 12: EOI (End of Infusion): number analyzed (Participants) | 3
  Week 12: EOI (End of Infusion) | 749 (215)
  Week 16: Pre-dose: number analyzed (Participants) | 3
  Week 16: Pre-dose | 201 (68.7)
  Week 16: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 20: Pre-dose: number analyzed (Participants) | 0
  Week 20: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 24: Pre-dose: number analyzed (Participants) | 0
  Week 24: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 28: Pre-dose: number analyzed (Participants) | 0
  Week 32: Pre-dose: number analyzed (Participants) | 0
  Week 32: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 36: Pre-dose: number analyzed (Participants) | 3
  Week 36: Pre-dose | 99.1 (171)
  Week 36: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 40: Pre-dose: number analyzed (Participants) | 0
  Week 40: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 44: Pre-dose: number analyzed (Participants) | 0
  Week 44: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 48: Pre-dose: number analyzed (Participants) | 0
  Week 48: EOI (End of Infusion): number analyzed (Participants) | 0
  Week 52: Pre-dose: number analyzed (Participants) | 0

18. Secondary Outcome: Concentration of Total Angiopoietin-like 3 (ANGPTL3) in Serum
Description: Concentration of total ANGPTL3 in serum by time were analyzed and reported.
Time Frame: as for outcome 17
Population: The total target analysis set included all treated participants who received any study drug and who had at least 1 non-missing post-dose total ANGPTL3 measurement following the first dose of study drug. Here, "number analyzed" signifies to participants evaluable for this outcome at given timepoints.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Evinacumab
Number analyzed (Participants) | 10 | 10
mg/L
  Week 0: Pre-Dose | 0.0930 (0.0225) | 0.0907 (0.0272)
  Week 0: EOI (End of Infusion) | 0.0826 (0.0180) | 0.211 (0.0362)
  Week 4: Pre-Dose: number analyzed (Participants) | 10 | 8
  Week 4: Pre-Dose | 0.0876 (0.0257) | 0.248 (0.105)
  Week 4: EOI (End of Infusion): number analyzed (Participants) | 10 | 8
  Week 4: EOI (End of Infusion) | 0.0828 (0.0260) | 0.306 (0.0992)
  Week 8: Pre-Dose: number analyzed (Participants) | 7 | 8
  Week 8: Pre-Dose | 0.0914 (0.0287) | 0.243 (0.0811)
  Week 8: EOI (End of Infusion): number analyzed (Participants) | 4 | 6
  Week 8: EOI (End of Infusion) | 0.0765 (0.0280) | 0.298 (0.0831)
  Week 12: Pre-Dose: number analyzed (Participants) | 5 | 5
  Week 12: Pre-Dose | 0.0767 (0.0121) | 0.281 (0.0851)
  Week 12: EOI (End of Infusion): number analyzed (Participants) | 3 | 3
  Week 12: EOI (End of Infusion) | 0.0699 (0.0106) | 0.322 (0.0672)
  Week 16: Pre-Dose: number analyzed (Participants) | 3 | 3
  Week 16: Pre-Dose | 0.0812 (0.0277) | 0.230 (0.0560)
  Week 16: EOI (End of Infusion): number analyzed (Participants) | 3 | 0
  Week 16: EOI (End of Infusion) | 0.0730 (0.0164) |
  Week 20: Pre-Dose: number analyzed (Participants) | 0 | 0
  Week 20: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 24: Pre-Dose: number analyzed (Participants) | 0 | 0
  Week 24: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 28: Pre-Dose: number analyzed (Participants) | 3 | 0
  Week 28: Pre-Dose | 0.0807 (0.0103) |
  Week 32: Pre-Dose: number analyzed (Participants) | 0 | 0
  Week 32: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 36: Pre-Dose: number analyzed (Participants) | 0 | 3
  Week 36: Pre-Dose |  | 0.162 (0.107)
  Week 36: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 40: Pre-Dose: number analyzed (Participants) | 0 | 0
  Week 40: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 44: Pre-Dose: number analyzed (Participants) | 0 | 0
  Week 44: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 48: Pre-Dose: number analyzed (Participants) | 0 | 0
  Week 48: EOI (End of Infusion): number analyzed (Participants) | 0 | 0
  Week 52: Pre-Dose: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to off drug follow-up (72 weeks)
Groups:
- Evinacumab 20 mg: Participants received evinacumab 20 mg/kg IV infusion Q4W starting from Day 1 up to 52 weeks.
Arm/Group | Placebo | Evinacumab 20 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/10 | 5/11
Other Adverse Events (participants affected / at risk) | 8/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Evinacumab 20 mg (N=11)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 2 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Evinacumab 20 mg (N=11)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 4 (5)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pedal pulse decreased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The sponsor terminated the study early due to enrollment issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT04863014/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT04863014/SAP_001.pdf